CLINICAL TRIAL: NCT04180579
Title: Safety and Tolerability of Lower Scalp Cooling Temperatures to Prevent Doxorubicin Plus Cyclophosphamide and Paclitaxel-induced Alopecia in Breast Cancer Patients
Brief Title: Safety of Lower Scalp Cooling Temperature to Prevent Hair Loss From Chemotherapy in Breast Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-277
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: alopecia; breast cancer; hair loss; chemotherapy induced alopecia; 19-277; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms; Alopecia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with Breast Cancer (Experimental): Any adult woman with a new diagnosis of breast cancer, Stage I-III
  Interventions: Device: PAXMAN Scalp Cooler

INTERVENTIONS:
Device: PAXMAN Scalp Cooler — Scalp cooling will occur with each dose of chemotherapy.

SUMMARY:
This study is being done to determine if using the Paxman Scalp Cooling System at temperatures lower than the current standard is a safe and tolerable approach to prevent hair loss in breast cancer patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* New diagnosis of breast cancer stage I-IV
* Planning to undergo neoadjuvant or adjuvant chemotherapy with curative intent
* Chemotherapy must be planned for at least 4 cycles of full-dose anthracycline plus cyclophosphamide followed by taxane based chemotherapy regimen:

  * Concurrent trastuzumab at standard doses is allowed
  * Concurrent pertuzumab at standard doses is allowed
  * Administration of chemotherapy on a dose dense schedule is allowed as clinically indicated
* For women of childbearing potential, a negative pregnancy test is needed within 7 days prior to study intervention, or whenever collected as per standard of care. For women who undergo fertility preservation or ovarian stimulation, a negative pregnancy test is not needed and eligibility due to positive pregnancy test will be determined by investigator discretion.

Exclusion Criteria:

* Any other concurrent malignancy including hematological malignancies (i.e. leukemia or lymphoma)
* Baseline alopecia (defined CTCAE v5.0 grade > 1)
* Subjects who are scheduled for bone marrow ablation chemotherapy
* Male gender
* Age >/= 75 years
* Personal history of migraines, cluster or tension headaches as defined as actual medical diagnosis by a physician and/or prescribed medications. If personal history of migraines was related to a past medical problem that is now resolved, subject may go on study at the discretion of the Principal Investigator.
* Subjects who have had prior chemotherapy
* Subjects who have had >/=1 previous chemotherapy exposure resulting in alopecia
* An existing history of scalp metastases or suspected presence of scalp metastasis
* Subjects with cold sensitivity, cryoglobulinemia, cryofibrinogenemia, or cold migraine pot-traumatic cold dystrophy
* Previously received, or scheduled to undergo skull irradiation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by CTCAE | Up to 44 weeks from the start of treatment
  Safety will be determined by toxicity assessment according to CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Shari Goldfarb, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org